CLINICAL TRIAL: NCT03102203
Title: Differentiation of Progression From Treatment Effects in High-Grade Gliomas: A Prospective Multicenter Clinical Trial With Multimodality MR Imaging
Brief Title: Differentiation of Progression From Treatment Effects in High-Grade Gliomas: A Clinical Trial With Multimodality MR Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Lu Guang Ming, Professor, Jinling Hospital, China
Other Study IDs: NanjingJH01
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the efficacy of multi-modality magnetic resonance quantitative parameters in evaluating the treatment effects of high-grade gliomas, and to provide new biomarkers for the establishment of new diagnostic criteria for the identification of true and pseudoprogression of high-grade gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high-grade gliomas confirmed by pathology and have not been treated with concurrent chemoradiotherapy;
2. Written informed consent is obtained.

Exclusion Criteria:

1. Patients not suitable for enhanced MRI scanning of patients;
2. Patients who have not finished follow-up concurrent chemoradiotherapy or MR scanning.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Eligibility module specifies the criteria for determining which people are (or are not) eligible to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Ktrans | baseline
  The volume transfer constant in dynamic contrast-enhanced MR Imaging
Ktrans | 3 months
  The volume transfer constant in dynamic contrast-enhanced MR Imaging
Ktrans | 10 months
  The volume transfer constant in dynamic contrast-enhanced MR Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ming Lu, Doctor, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China